CLINICAL TRIAL: NCT02823054
Title: One-lung Ventilation During Internal Thoracic Artery Grafting in Cardiac Surgery
Acronym: VUPPAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI2015_843_0013
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Bypass
Keywords: elective surgery; CABG; One-lung ventilation; EZ Blockers; pleural effusion
MeSH Terms: conditions — Pleural Effusion

ARMS (2):
- Standard group (No Intervention): bi lung ventilation usual practice
- EZ-Blocker group (Experimental): one lung ventilation 'EZ-Blocker'
  Interventions: Device: EZ-Blocker

INTERVENTIONS:
Device: EZ-Blocker — the Blocker group, the EZ-Blocker will be set up after anesthesia induction and standard orotracheal intubation to allow lung exclusion during homolateral internal thoracic artery sampling, and thus a one-lung ventilation. This material will be removed at the end of surgical surgery.
  Arms: EZ-Blocker group

SUMMARY:
Coronary artery bypass grafting is a current cardiac surgery. Internal thoracic artery is usually taking to restore coronary revascularization, and its dissection can lead to accidental or voluntary pleural effusions. Respiratory complications are frequent, due to the drainage required. In this study, the investigators propose one-lung ventilation to facilitate artery grafting and surgical procedure. The investigators will include all adult patients with elective coronary artery bypass surgery (CABG) by internal thoracic artery, in a prospective, controlled, randomized and monocentric study. The main objective is to demonstrate that one-lung ventilation using EZ-Blocker can reduce pleural effusion defined by presence of drainage and/or pneumothorax on X-ray chest in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* elective CABG surgery with internal thoracic artery, with patient consent.
* Patient who have french social security

Exclusion Criteria:

* Cardiac or thoracic past-history
* polyurethane allergy
* guardianship patient
* endotracheal intern diameter too small to allow the EZ-Blocker introduction or the fiberscope
* use of LASER immediately near the EZ-Blocker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Pleural effusions after coronary artery bypass graft surgery | Day 0
  quantifying the number of thoracic drains (0, 1 or 2), as accidental or voluntary pleural effusion
absence of pneumothorax | Day 0
  verify the absence of pneumothorax to X-ray chest ( not drained pleural effusion).

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu GUILBART, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France